CLINICAL TRIAL: NCT01159080
Title: Organ Function Preservation by the Combination Treatment of the optImuM Dose of calcineUrin Inhibitor and Mycophenolate Sodium in Kidney Recipients: OPTIMUM Study
Brief Title: Treatment of the optImuM Dose of calcineUrin Inhibitor and Mycophenolate Sodium in Kidney Recipients
Acronym: OPTIMUM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Seoul National University Hospital (Other); Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Su-Kil Park, Professor, Department of medicine, ASAN Medical CENTER, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CERL080AKR07T; CERL080AKR07T (Other Grant/Funding Number: NORVATIS)
Record Dates: First submitted 2010-07-06; First posted 2010-07-09 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Kidney Transplantation
Keywords: immunosuppression control in kidney transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- routine dose tacrolimus and less myfortic (Active Comparator)
  Interventions: Drug: routine dose tacrolimus and less myfortic
- reduced dose tacrolimus and conventional myfortic (Experimental)
  Interventions: Drug: reduced dose tacrolimus and conventional myfortic

INTERVENTIONS:
Drug: routine dose tacrolimus and less myfortic — oral regular dose of tacrolimus + less dose of myfortic trough level of tacrolimus will be 5-10 ng/mL and oral myfortic dose will be 180-360 mg twice a day
  Arms: routine dose tacrolimus and less myfortic
Drug: reduced dose tacrolimus and conventional myfortic — low dose of tacrolimus + maximum dose of myfortic target trough level of tacrolimus should be reduced to 2-5 ng/mL for 3 months after randomization and oral MPS dose increased to 540-720mg twice a day
  Arms: reduced dose tacrolimus and conventional myfortic

SUMMARY:
To clarify that tacrolimus-sparing regimen with minimal tacrolimus dose together with mycophenolate sodium dose increment will preserve renal allograft function without rising adverse effects

Primary endpoints:

1. estimated GFR (MDRD equation) 12 months after randomization
2. estimated GFR change from randomization to end of the study (calculated by MDRD equation and Nankivell equation)

ELIGIBILITY:
<Inclusion criteria>

1. The patients between the ages of 20 and 75 years who received kidney transplantation one to five years prior to the study.
2. Taking tacrolimus and corticosteroid, with or without additional purine synthesis inhibitor within the recent 3 months
3. Patients with serum creatinine (sCr) level ≤ 2.0 mg/dL and variation of sCr < 30% for recent 3 months
4. Patients with urine proteinuria/creatinine ratio (PCR) ≤ 1 g/g, or 24 hour urine protein ≤ 1g/day for recent 3 months
5. Patients who provided informed consent.

<Exclusion criteria>

1. Patients who received combined non-renal transplantation, multiple kidney transplantation or re-transplantation
2. Patients whose graft from non-heart beating cadaveric donor
3. graft from HLA-identical living related donor
4. ABO blood group incompatible donor or HLA desensitized recipients
5. Patients with hypersensitivity history to mycophenolate sodium, mycophenolate acid, or mycophenolate mofetil, or to any other excipients
6. Patients with hypoxanthin e-guanine phosphoribosyl-transferase such as Lesch-Nyhan syndrome and Kelley-Seegmiller syndrome
7. Patients with history of disease which could affect absorption of study medication (e.g. diabetic gastropathy, previous gastrectomy)
8. Patients with positive serologic test results, in recipient or donor, for human immunodeficiency virus, hepatitis B or C virus
9. Patients with liver function test abnormality (alanine aminotransferase, aspartate aminotransferase, or total bilirubin > 3 times from upper normal limit), neutropenia (absolute neutrophil count < 1,500/uL or white blood cell count < 2,500/uL), or thrombocytopenia (platelet < 75,000)
10. Patients with history of cancer within 5 years, except for successfully treated localized non-melanocytic skin cancer
11. Patients who were either pregnant, lactating, planning to become pregnant in the next 12 months
12. Patients who taken medicine from other trial within 30 days.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2010-04-01 (Actual); Primary Completion 2016-10-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
estimated GFR (MDRD equation)12 months after randomization | 12 months after randomization

SECONDARY OUTCOMES:
Urine protein excretion | 12 months after randomization
  24hr urine collection or urine protein/creatinine ratio
graft survival | 12 month after randomization
  12 month graft survival
follow-up loss | From randomization to 12 months after randomization
  frequency of follow-up loss
Allograft biopsy | From randomization to 12 months after randomization
  number of performed allograft biopsy performed
Treated or biopsy proven acute rejection | From randomization to 12 months after randomization
estimated GFR change from randomization to end of the study | 12 months after randomization
  calculated by MDRD equation and Nankivell equation

CONTACTS AND LOCATIONS:
Overall Officials: Su-Kil Park, MD,PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Asan Medical Center, South Korea

REFERENCES:
- [Derived] Park S, Kim YS, Lee J, Huh W, Yang CW, Kim YL, Kim YH, Kim JK, Oh CK, Park SK. Reduced Tacrolimus Trough Level Is Reflected by Estimated Glomerular Filtration Rate (eGFR) Changes in Stable Renal Transplantation Recipients: Results of the OPTIMUM Phase 3 Randomized Controlled Study. Ann Transplant. 2018 Jun 12;23:401-411. doi: 10.12659/AOT.909036. PMID 29891834